CLINICAL TRIAL: NCT05646641
Title: Does Strength Training in Fibromyalgia Affect Balance, Neuromuscular Performance and Symptoms? A 12 Week of a Randomized Controlled Trial
Brief Title: Strength Training in Fibromyalgia on Balance, Neuromuscular Performance and Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria Luiza Laurentino de Albuquerque, Principal Investigator, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2834
Record Dates: First submitted 2022-11-29; First posted 2022-12-12 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 8 weeks of strength training.
  Interventions: Other: Strength exercise
- Control (No Intervention): Maintain their usual medical treatment and daily routines

INTERVENTIONS:
Other: Strength exercise — The protocol consists of 8 weeks of training, consisting of 16 sessions of 50 minutes, twice a week on alternate days.
  Arms: Exercise

SUMMARY:
The purpose of this study is verify the effects of a 8 weeks strength training, on balance, neuromuscular performance and symptomatology of fibromyalgia.

DETAILED DESCRIPTION:
Thirty participants will be recruited. Volunteers will be randomly assigned to the control group or experimental group. Before the training period, symptoms, balance and neuromuscular performance will be assessed. Participants in the experimental group will perform strength training twice a week (50 min each) for eight weeks. Then, four weeks of detraining will be completed.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of fibromyalgia according to the American College of Rheumatology criteria
* at least 18 years old

Exclusion Criteria:

* severe comorbidity or any other type of condition that negatively influences participation in the training program
* cognitive disorders
* heart problems
* surgeries or fractures in the last 6 months
* regular practice of physical exercises in the least 3 months before program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Balance | Change from Baseline balance at week 9
  Force plate
Balance | Change from Baseline balance at week 12
  Force plate
Balance | Change from week 9 balance at week 12
  Force plate
Neuromuscular performance | Change from Baseline neuromuscular performance at week 9
  Optical measurement system consisting of two transmitting and receiving cells to assess vertical jump and medicine ball to assess strength of the upper limbs.
Neuromuscular performance | Change from Baseline neuromuscular performance at week 12
  Optical measurement system consisting of two transmitting and receiving cells to assess vertical jump and medicine ball to assess strength of the upper limbs.
Neuromuscular performance | Change from week 9 neuromuscular performance at week 12
  Optical measurement system consisting of two transmitting and receiving cells to assess vertical jump and medicine ball to assess strength of the upper limbs.

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire | Baseline, week 9, week 12
  Questionnaire to ccess information on the functional capacity and health status of individuals with fibromyalgia. Composed of 20 questions. , the values vary from 0 to 100, in which the higher the value, the greater the impact of fibromyalgia.
Pain intensity | baseline and everyday until the week 12
  Visual Analogue Scale (VAS). The scoring range will be from 0 to 100, in which the higher the value, the greater the intensity. During non-presencial days, participants will respond daily the intensity with a cell phone application developed for this purpose.
Anxiety | baseline and everyday until the week 12
  Visual Analogue Scale (VAS). The scoring range will be from 0 to 100, in which the higher the value, the greater the intensity. During non-presencial days, participants will respond daily the intensity with a cell phone application developed for this purpose.
Quality of sleep | baseline and everyday until the week 12
  Visual Analogue Scale (VAS). The scoring range will be from 0 to 100, in which the higher the value, the greater the intensity. During non-presencial days, participants will respond daily the intensity with a cell phone application developed for this purpose.
Fatigue | baseline and everyday until the week 12
  Visual Analogue Scale (VAS). The scoring range will be from 0 to 100, in which the higher the value, the greater the intensity. During non-presencial days, participants will respond daily the intensity with a cell phone application developed for this purpose.
Mood state | baseline and everyday until the week 12
  Visual Analogue Scale (VAS). The scoring range will be from 0 to 100, in which the higher the value, the greater the intensity. During non-presencial days, participants will respond daily the intensity with a cell phone application developed for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Study Director — University of Beira Interior
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albuquerque MLL, Monteiro D, Alvarez MC, Vilarino GT, Andrade A, Neiva HP. Effects of strength training in fibromyalgia on balance, neuromuscular performance, and symptomatic analysis: a 12-week study protocol. Front Neurol. 2023 Apr 28;14:1149268. doi: 10.3389/fneur.2023.1149268. eCollection 2023. PMID 37188309